CLINICAL TRIAL: NCT05676866
Title: Evaluation of Targeted Axillary Lymph Nodes Dissection in Node Positive Breast Cancer Patients Post Neo Adjuvant Therapy
Brief Title: Evaluation of Targeted Axillary Lymph Node Dissection in Node Positive Breast Cancer Patients Post Neo Adjuvant Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Abdelnasser Mahmoud Ali, Resident doctor /Omar abdelnasser Mahmoud, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Targeted axillary dissection
Record Dates: First submitted 2023-01-02; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Node-positive Breast Cancer

STUDY DESIGN:
Intervention Model Description: Node positive breast cancer patients post neo adjuvant therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer patients with positive axillary nodes (Experimental): Female with invasive breast cancer with axillary metastasis , who recieve neo adjuvant therapy with complete axillary response
  Interventions: Procedure: Targeted axillary lymph node dissection

INTERVENTIONS:
Procedure: Targeted axillary lymph node dissection — Targeted axillary lymph node dissection is done by marking suspicious node with metallic clip prior to neo adjuvant therapy ,then neo adjuvant therapy is given and after complete axillary response (proved by radiological and clinical examination) , targeted axillary lymph node dissection of clipped node is done along with sentinel lymph node dissection

SUMMARY:
evaluation of targeted axillary lymph node dissection in node positive breast cancer patients post neo adjuvant therapy

DETAILED DESCRIPTION:
Targeted axillary dissection (TAD) is a novel technique in the field of surgical oncology. During TAD, patients with node-positive breast cancer who clinically responded to neoadjuvant chemotherapy undergo resection of a previously proven metastatic node together with sentinel lymph node dissection (SLND).

Compared to sentinel lymph node dissection (SLND), axillary lymph node dissection [ALND] is associated with increased morbidity, higher rates of lymphedema, paraesthesia, sensory loss in the arm, and impairment in shoulder function. Patients undergoing SLND have fewer infections and a better quality of life, so axillary dissection has been largely replaced by SLND in early-stage breast cancer.

Targeted axillary dissection (TAD) is an innovative surgical procedure that emerged in an attempt to further decrease the false negative results of SLND.

Breast cancer patients suitable for neoadjuvant systemic therapy [NAST] with node-positive disease (N1,N2) were assessed by the multi-disciplinary team and if potentially eligible for TAD, a metallic marker[clip] is inserted in the suspicious node prior to neoadjuvant therapy.

The procedure is performed together with SLND using a single-tracer technique. Towards the end of NAST, a progress ultrasound and mammogram are performed to assess the breast and axillary response, Clip position within node is confirmed.

A standard surgical approach for sentinel lymph node dissection [SLND] is used for TAD, Patent blue dye is administered intraoperatively. dissection down to the localized node is performed. node contained the clip is subsequently sent for histology. Any residual sentinel nodes or palpable abnormal nodes are excised and examined separately.

ELIGIBILITY:
Inclusion Criteria:

1. females with invasive breast cancer with axillary metastasis, staging of n1: n2
2. complete axillary response to neoadjuvant therapy by clinical examination and imaging

Exclusion Criteria:

* 1. breast cancer patients who are not candidate for neoadjuvant chemotherapy 2. breast cancer patients with positive axillary node post neoadjuvant chemotherapy 3. breast cancer patients with distant metastasis 4. patients with axillary lymph node metastasis from another primary tumour [not breast cancer]

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female patients with breast cancer and axillary metastasis
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation the sensitivity of targeted axillary lymph node dissection in node positive breast cancer patients | 3 monthes
Comparing sensetivity of targeted axillary dissection with traditional SLND | 3 monthes

SECONDARY OUTCOMES:
Post operative complications: number of patients with arm lymphedema and sensory loss | 3 monthes

REFERENCES:
- See also: The Feasibility and Accuracy of Sentinel Lymph Node Biopsy in Initially Clinically Node-Negative Breast Cancer after Neoadjuvant Chemotherapy: A Systematic Review and Meta-Analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5015960/
- See also: Targeted Axillary Dissection in Node-Positive Breast Cancer: A Retrospective Study and Cost Analysis — https://www.cureus.com/articles/44726-targeted-axillary-dissection-in-node-positive-breast-cancer-a-retrospective-study-and-cost-analysis
- See also: Improved Model for Predicting Axillary Response to Neoadjuvant Chemotherapy in Patients with Clinically Node-Positive Breast Cancer — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5743998/
- See also: Feasibility and Accuracy of Sentinel Lymph Node Biopsy in Clinically Node-Positive Breast Cancer after Neoadjuvant Chemotherapy: A Meta-Analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4161347/
- See also: Comprehensive Axillary Evaluation in Neoadjuvant Chemotherapy Patients With Ultrasonography and Sentinel Lymph Node Biopsy — https://link.springer.com/article/10.1245/ASO.2005.09.007